CLINICAL TRIAL: NCT00135694
Title: A Phase II Trial to Assess the Safety of Immunosuppression Withdrawal in Liver Transplant Recipients
Brief Title: Gradual Withdrawal of Immune System Suppressing Drugs in Patients Receiving a Liver Transplant
Acronym: A-WISH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN030ST
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C; Hepatitis C, Chronic; Nonimmune Nonviral Causes of Liver Failure
Keywords: hepatitis; hepatitis C; HCV; liver; liver disease; liver transplant; liver transplantation; transplant; hepatic; hepatic transplantation; immunosuppression; rejection
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Hepatitis; Liver Diseases; Rejection, Psychology | interventions — Liver Transplantation; Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunosuppression Withdrawal (Experimental): Subjects may randomize to this group at 12 to 24 months after transplantation. This is followed by tapered withdrawal of calcineurin inhibitor-based immunosuppression therapy over the course of 1 year.
  Interventions: Drug: calcineurin inhibitor-based immunosuppression; Procedure: liver transplant; Drug: corticosteroids; Other: immunosuppression withdrawal
- Immunosuppression Maintenance (Active Comparator): Liver transplant, followed by maintenance doses of continuous calcineurin inhibitor-based immunosuppression therapy.
  Interventions: Drug: calcineurin inhibitor-based immunosuppression; Procedure: liver transplant; Drug: corticosteroids

INTERVENTIONS:
Drug: calcineurin inhibitor-based immunosuppression — May be cyclosporine, mycophenolate mofetil, or tacrolimus
Procedure: liver transplant — Occurs at study entry
  Other Names: liver transplantation
Drug: corticosteroids — 3-month course of corticosteroids
  Other Names: prednisone
Other: immunosuppression withdrawal — One year after transplantation, participants eligible for withdrawal are randomly assigned in a 4 to 1 ratio to immunosuppression withdrawal or to maintenance.
  Arms: Immunosuppression Withdrawal

SUMMARY:
In order to prevent organ rejection, patients receiving liver transplants currently require life-long treatment with immune system-suppressing medications to prevent the rejection of the transplanted liver. However, these medications can cause long-term side effects, such as infection, kidney problems, diabetes, and cancer. In patients infected with hepatitis C virus (HCV), these medications may increase the risk of HCV infection in the transplanted liver. The purpose of this study is to determine whether a slow withdrawal of immune system-suppressing medications is safe in two groups of subjects: those who receive a liver transplant due to HCV, and those who receive a liver transplant due to non-immune, non-viral causes of liver failure. The study will also look at whether slow withdrawal will help reduce the long-term side effects of immune system-suppressing medications and decrease the chance for HCV infection of the new liver in transplant patients with HCV.

DETAILED DESCRIPTION:
This is a prospective multicenter, open-label, randomized trial in which individuals with liver failure due to hepatitis C or to nonimmune nonviral causes undergo liver transplantation and receive immunosuppression with a calcineurin inhibitor and corticosteroids. Corticosteroids are tapered in the 3 months after transplantation and the calcineurin inhibitor is continued. Participants are regularly assessed for evidence of allograft rejection. One year after transplantation, participants eligible for withdrawal are randomly assigned in a 4 to 1 ratio to immunosuppression withdrawal or to maintenance. Participants assigned to withdrawal undergo a scheduled taper over approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. Necessity for liver transplant.
3. For females of childbearing potential: a negative pregnancy test at study entry and agreement to use approved methods of birth control for the duration of their participation.
4. Ability to provide informed consent.
5. Availability of donor specimen(s).
6. For individuals with hepatitis C infection, presence of hepatitis genomes in blood.

Exclusion Criteria:

1. Previous transplant.
2. Multiorgan or split liver transplant other than with a right trisegment.
3. Living donor transplant.
4. Donor liver from a donor positive for antibody against hepatitis C.
5. Donor liver from a non-heart-beating donor.
6. Liver failure due to autoimmune disease.
7. Fulminant liver failure.
8. Hepatitis B infection as defined by the presence of HbSAg or hepatitis-C infection with a genome other than genome 1.
9. Stage III or higher hepatocellular cancer.
10. History of malignancy except hepatocellular cancer, adequately treated in situ cervical carcinoma,adequately treated basal or squamous cell carcinoma of skin, or other cancer judged to have a 5-year risk of recurrence less than 10%.
11. Active systemic infection at the time of transplantation.
12. Clinically significant chronic renal disease.
13. Clinically significant cardiovascular or cerebrovascular disease.
14. Infection with human immunodeficiency virus.
15. Any investigational drug received within 6 weeks of study entry or any investigational vaccine received at any time.
16. Hypersensitivity to tacrolimus.
17. Unwillingness or inability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2005-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Shaked, MD, PhD, Study Chair — University of Pennsylvania
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor University, Dallas, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Shaked A, DesMarais MR, Kopetskie H, Feng S, Punch JD, Levitsky J, Reyes J, Klintmalm GB, Demetris AJ, Burrell BE, Priore A, Bridges ND, Sayre PH. Outcomes of immunosuppression minimization and withdrawal early after liver transplantation. Am J Transplant. 2019 May;19(5):1397-1409. doi: 10.1111/ajt.15205. Epub 2018 Dec 31. PMID 30506630
- [Derived] Muthukumar T, Akat KM, Yang H, Schwartz JE, Li C, Bang H, Ben-Dov IZ, Lee JR, Ikle D, Demetris AJ, Tuschl T, Suthanthiran M. Serum MicroRNA Transcriptomics and Acute Rejection or Recurrent Hepatitis C Virus in Human Liver Allograft Recipients: A Pilot Study. Transplantation. 2022 Apr 1;106(4):806-820. doi: 10.1097/TP.0000000000003815. PMID 33979314
- See also: National Institute of Allergy and Infectious Diseases website — https://www.niaid.nih.gov/
- See also: Click here for the Immune Tolerance Network website — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with liver failure due to hepatitis C infection or non-immune, non-viral causes were enrolled between October 2005 and April 2011.
Pre-assignment Details: Participants 12-24 months post-transplant, stable on immunosuppression monotherapy for at least 3 months prior to random assignment, with stage 2 or less fibrosis on the Ishak scale, adequate hepatic and renal function, and no biopsy-proven rejection were randomized between November 2006 and December 2012.
Groups:
- Terminated Prior to Randomization: Subjects enrolled and transplanted into the trial but not eligible for randomization.
- Randomized to Immunosuppression Withdrawal: Subjects enrolled and transplanted into the trial and followed for at least one year and eligible for random assignment and randomized to immunosuppression withdrawal.
- Randomized to Immunosuppression Maintenance: Subjects enrolled and transplanted into the trial and followed for at least one year and eligible for random assignment and randomized to immunosuppression maintenance.
Period: Overall Study
Arm/Group | Terminated Prior to Randomization | Randomized to Immunosuppression Withdrawal | Randomized to Immunosuppression Maintenance
Started | 180 | 77 | 18
Completed | 0 (Subjects were assessed as ineligible for random assignment and subsequently terminated per protocol.) | 56 | 11
Not Completed | 180 | 21 | 7
Not completed — Adverse Event | 17 | 4 | 0
Not completed — Death | 14 | 1 | 2
Not completed — Lost to Follow-up | 8 | 7 | 1
Not completed — Withdrawal by Subject | 41 | 7 | 4
Not completed — Protocol Violation | 19 | 1 | 0
Not completed — Hepatitis C related reasons | 39 | 1 | 0
Not completed — Ineligible for Random assignment | 42 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled sample (subjects transplanted in the study)
Groups:
- Total: Total of all reporting groups
Arm/Group | Terminated Prior to Randomization | Randomized to Immunosuppression Withdrawal | Randomized to Immunosuppression Maintenance | Total
Number analyzed (Participants) | 180 | 77 | 18 | 275
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 161 | 68 | 13 | 242
  >=65 years | 19 | 9 | 5 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (7.83) | 54.3 (9.92) | 57.4 (7.70) | 55.3 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 14 | 5 | 72
  Male | 127 | 63 | 13 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 3 | 24
  Not Hispanic or Latino | 167 | 66 | 15 | 248
  Unknown or Not Reported | 3 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 22 | 7 | 0 | 29
  White | 153 | 66 | 17 | 236
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 180 | 77 | 18 | 275
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] — The latest creatinine value collected at the screening or baseline visit prior to transplant was used for this measure. The test measures kidney function. According to Harrison's Principles of Internal Medicine, normal results are 0.6 to 1.2 mg/dL for men and 0.5 to 0.9 mg/dL for women. Abnormal kidney function results in increased levels of serum creatinine.
  mg/dL | 1.5 (1.18) | 1.3 (0.65) | 1.1 (0.68) | 1.4 (1.04)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Complications Usually Attributed to Immunosuppression
Description: This is a composite endpoint comprising clinical complications related to immunosuppression and is defined as the occurrence of any of the following: death or graft loss, grade 4 secondary malignancy (graded by Common Terminology Criteria for Adverse Events [CTCAE] version 3.0), grade 4 opportunistic infection (graded by CTCAE version 3.0), stage 3 or higher fibrosis, or decrease in renal function. Decrease in renal function is defined as: a) the estimated glomerular filtration rate (eGFR) using creatinine obtained prior to and closest to randomization will be considered the baseline and will be compared to the eGFR using creatinine obtained at 24 months +/- 3 months after randomization; b) for those with a baseline eGFR 30-90 ml per min per 1.73 meter-squared, a 25% decrease in eGFR; c) for those with a baseline eGFR greater than 90 ml per min per 1.73 meter-squared, a 25% decrease in eGFR and a decrease in eGFR to less than 90 ml per min per 1.73 meter-squared.
Time Frame: Randomization to 2 years post-randomization
Population: Evaluable randomized subjects having a targeted event and/or having available data for calculation of eGFR
Measure: Number; unit: participants
Arm/Group | Randomized to Immunosuppression Withdrawal | Randomized to Immunosuppression Maintenance
Number analyzed (Participants) | 66 | 13
participants | 12 | 4
Statistical Analysis 1: Comparison: Randomized to Immunosuppression Withdrawal vs Randomized to Immunosuppression Maintenance; Test type: Superiority or Other; Risk Difference (RD) = -13, 90% CI 2-sided [-35 to 10]

2. Secondary Outcome: Number of Participants Who Qualify for Random Assignment
Time Frame: One to two years post-transplantation
Population: All subjects transplanted
Measure: Number; unit: participants
Groups:
- All Enrolled: Subjects who underwent liver transplantation in the trial.
Arm/Group | All Enrolled
Number analyzed (Participants) | 275
participants | 95

3. Secondary Outcome: Number of Participants Who Successfully Stop Taking Immunosuppression for at Least 6 Months
Time Frame: Randomization until study completion or participant termination (up to six years post-transplant)
Population: Participants randomized to immunosuppression withdrawal
Measure: Number; unit: participants
Arm/Group | Randomized to Immunosuppression Withdrawal
Number analyzed (Participants) | 77
participants | 12

4. Secondary Outcome: Immunosuppression-free Duration
Description: Time (in days) from withdrawing off of all immunosuppressive drugs to re-starting immunosuppression or study termination/completion.
Time Frame: Discontinuation of all immunosuppression to end of trial participation or to time of restarting immunosuppression, whichever came first, assessed up to two years
Population: Participants randomized to immunosuppression withdrawal who completed withdrawal and discontinued all immunosuppression
Measure: Mean (Full Range); unit: Days
Arm/Group | Randomized to Immunosuppression Withdrawal
Number analyzed (Participants) | 14
Days | 555.2 [36 to 790]

5. Secondary Outcome: Number of Hepatitis C Infected Participants With Progression of Hepatitis C Related Liver Disease, Defined as Stage 4 or Higher Fibrosis on the Ishak Scale
Description: Number of subjects with a biopsy showing stage 4 fibrosis or higher on the Ishak scale. Stage 4 represents at least 13.7% fibrosis measurement with a description of fibrous expansion of portal areas with marked bridging (P-P) as well as portal to central (P-C). Stage 5 is marked bridging (P-P and/or P-C), with occasional nodules (incomplete cirrhosis) and stage 6 is cirrhosis, probable or definite.
Time Frame: Randomization to 2 years post-randomization.
Population: Hepatitis C infected participants randomized.
Measure: Number; unit: participants
Arm/Group | Randomized to Immunosuppression Withdrawal | Randomized to Immunosuppression Maintenance
Number analyzed (Participants) | 30 | 7
participants | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing Graft Loss or Death
Description: Number of participants with graft loss or death. Graft loss is defined as subject death or re-transplantation.
Time Frame: Randomization to 2 years post-randomization.
Population: Randomized participants (intent-to-treat sample)
Measure: Number; unit: participants
Arm/Group | Randomized to Immunosuppression Withdrawal | Randomized to Immunosuppression Maintenance
Number analyzed (Participants) | 77 | 18
participants | 1 | 0

7. Secondary Outcome: Total Immunosuppression From Month 21 to Month 24 Post-randomization
Description: Daily immunosuppression score in units per day averaged over the 3-month period from Month 21 to Month 24 post-randomization. Daily doses were assigned a score of 1 unit as follows: tacrolimus 1 mg, cyclosporine 100 mg, Sirolimus 1 mg, mycophenolate mofetil 1000 mg, Mycophenolic acid 720 mg, azathioprine 50 mg, and prednisone 5 mg. Any antibody use equaled 20 units. Unit scores based on Vasudev (Vasudev B, Hariharan S, Hussain SA, Zhu YR, Bresnahan BA et al. BK virus nephritis: risk factors, timing, and outcome in renal transplant recipients. Kidney Int. 2005; 8(4):1834-1839.)
Time Frame: Month 21 to Month 24 post-randomization
Population: Randomized participants still being followed 24 months post-randomization.
Measure: Mean (Full Range); unit: units per day
Arm/Group | Randomized to Immunosuppression Withdrawal | Randomized to Immunosuppression Maintenance
Number analyzed (Participants) | 64 | 13
units per day | 2.8 [0.0 to 10.0] | 3.7 [1.5 to 8.0]
Statistical Analysis 1: Comparison: Randomized to Immunosuppression Withdrawal vs Randomized to Immunosuppression Maintenance; Test type: Superiority or Other; p = 0.0183, ANCOVA; Adjusted for immunosuppression dose the subject was receiving at the time of randomization

8. Secondary Outcome: Total Burden of Immunosuppression From Random Assignment to Month 24
Description: Total immunosuppression score in units taken as the sum of units per day over the 2-year period from randomization to Month 24 post-randomization. Daily doses were assigned a score of 1 unit as follows: tacrolimus 1 mg, cyclosporine 100 mg, Sirolimus 1 mg, mycophenolate mofetil 1000 mg, Mycophenolic acid 720 mg, azathioprine 50 mg, and prednisone 5 mg. Any antibody use equaled 20 units. Unit scores based on Vasudev (Vasudev B, Hariharan S, Hussain SA, Zhu YR, Bresnahan BA et al. BK virus nephritis: risk factors, timing, and outcome in renal transplant recipients. Kidney Int. 2005; 8(4):1834-1839.).
Time Frame: Randomization to Month 24 post-randomization
Population: Randomized participants still being followed 24 months post-randomization.
Measure: Mean (Full Range); unit: units
Arm/Group | Randomized to Immunosuppression Withdrawal | Randomized to Immunosuppression Maintenance
Number analyzed (Participants) | 64 | 13
units | 2198.5 [255 to 4604] | 2708.4 [1126 to 6853]
Statistical Analysis 1: Comparison: Randomized to Immunosuppression Withdrawal vs Randomized to Immunosuppression Maintenance; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted for immunosuppression dose the subject was receiving at the time of randomization

ADVERSE EVENTS:
Time Frame: Enrollment through end of study (up to 7 years)
Arm/Group | Terminated Prior to Randomization | Randomized to Immunosuppression Withdrawal | Randomized to Immunosuppression Maintenance
Serious Adverse Events (participants affected / at risk) | 89/180 | 9/18 | 54/77
Other Adverse Events (participants affected / at risk) | 155/180 | 18/18 | 76/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terminated Prior to Randomization (N=180) | Randomized to Immunosuppression Withdrawal (N=18) | Randomized to Immunosuppression Maintenance (N=77)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 0 (0) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 4 (6) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Intestinal strangulation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peritoneal effusion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia obstructive (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 0 (0) | 4 (4)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 4 (4)
Cholangitis (Hepatobiliary disorders) | 4 (5) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic artery stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 26 (28) | 1 (1) | 21 (25)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cryptococcosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 7 (7) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Perihepatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 8 (8) | 2 (2) | 2 (2)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Graft dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 6 (6)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 7 (7) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 4 (4) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 0 (0) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (11) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Central pontine myelinolysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 5 (5) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 5 (5) | 0 (0) | 3 (5)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Treatment noncompliance (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Haematoma evacuation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Medical device change (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Small intestinal resection (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terminated Prior to Randomization (N=180) | Randomized to Immunosuppression Withdrawal (N=18) | Randomized to Immunosuppression Maintenance (N=77)
Anaemia (Blood and lymphatic system disorders) | 27 (37) | 3 (3) | 11 (14)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 2 (2) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular icterus (Eye disorders) | 6 (6) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 1 (1) | 3 (3)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 0 (0) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4)
Ascites (Gastrointestinal disorders) | 13 (15) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (7) | 0 (0) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 25 (28) | 2 (2) | 13 (18)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (5)
Nausea (Gastrointestinal disorders) | 11 (12) | 2 (2) | 10 (13)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 6 (6) | 0 (0) | 9 (11)
Asthenia (General disorders) | 4 (4) | 1 (1) | 2 (2)
Fatigue (General disorders) | 8 (9) | 0 (0) | 8 (9)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 5 (7)
Oedema (General disorders) | 12 (14) | 0 (0) | 5 (5)
Oedema peripheral (General disorders) | 43 (45) | 4 (4) | 16 (18)
Pyrexia (General disorders) | 15 (17) | 1 (1) | 13 (17)
Bile duct stenosis (Hepatobiliary disorders) | 8 (8) | 0 (0) | 6 (6)
Biloma (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 18 (18) | 2 (2) | 15 (15)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 5 (5)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 7 (7)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 4 (6)
Hepatitis C (Infections and infestations) | 35 (35) | 2 (2) | 16 (16)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (5)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0) | 5 (5)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 8 (11)
Urinary tract infection (Infections and infestations) | 14 (16) | 0 (0) | 10 (22)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 4 (4)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Incision site complication (Injury, poisoning and procedural complications) | 8 (8) | 1 (1) | 6 (6)
Incision site pain (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 6 (7)
Incisional hernia (Injury, poisoning and procedural complications) | 6 (6) | 3 (3) | 2 (2)
Post procedural bile leak (Injury, poisoning and procedural complications) | 14 (15) | 2 (2) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 6 (10)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 5 (9)
Blood alkaline phosphatase increased (Investigations) | 3 (4) | 1 (1) | 6 (7)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1) | 3 (5)
Blood creatinine increased (Investigations) | 8 (8) | 1 (1) | 8 (8)
Blood glucose increased (Investigations) | 4 (4) | 1 (1) | 4 (4)
Breath sounds abnormal (Investigations) | 11 (12) | 3 (3) | 11 (12)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 1 (1) | 5 (7)
Haematocrit decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 3 (3) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 7 (7) | 0 (0) | 9 (9)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Liver function test abnormal (Investigations) | 14 (14) | 3 (4) | 25 (32)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 29 (29) | 2 (3) | 20 (20)
Gout (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 19 (19) | 0 (0) | 15 (17)
Hyperkalaemia (Metabolism and nutrition disorders) | 28 (35) | 3 (3) | 23 (28)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 (14) | 2 (2) | 13 (14)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 10 (10)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 4 (4)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 13 (13) | 0 (0) | 11 (15)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 1 (1) | 5 (5)
Tremor (Nervous system disorders) | 11 (12) | 2 (2) | 9 (13)
Confusional state (Psychiatric disorders) | 10 (10) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 6 (6) | 3 (5) | 5 (5)
Insomnia (Psychiatric disorders) | 6 (6) | 0 (0) | 6 (7)
Renal failure (Renal and urinary disorders) | 27 (27) | 3 (3) | 15 (16)
Renal failure acute (Renal and urinary disorders) | 12 (13) | 0 (0) | 4 (4)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 1 (1) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 1 (1) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (2) | 4 (5)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Finger amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 12 (12) | 2 (2) | 9 (9)
Hypotension (Vascular disorders) | 5 (5) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No